CLINICAL TRIAL: NCT06719297
Title: Cognitive Integrated Motor Training to Improve Gait and Balance and Reduce Falls in Older Adults With Mild Cognitive Impairment
Brief Title: Cognitive Integrated Motor Training (CM) to Improve Gait and Balance and Reduce Falls in Older Adults With Mild Cognitive Impairment
Acronym: CM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Rutgers University (Other); New Jersey Institute of Technology (Other)
Responsible Party: Principal Investigator, Kiran Karunakaran, Research Scientist, Principal Investigator, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-1276-24; 90IFRE0092 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2024-11-18; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment
Keywords: older adults, mild cognitive impairment, gait, balance
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized cognitive-sensorimotor VR/MR training (Experimental): Thinking task integrated walking and balance training program
  Interventions: Other: Personalized cognitive-sensorimotor VR/MR training
- Standard of Care (Active Comparator): Standard walking and balance training
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Personalized cognitive-sensorimotor VR/MR training — Thinking task integrated walking and balance training program
  Arms: Personalized cognitive-sensorimotor VR/MR training
Other: Standard of Care — Standard walking and balance training
  Arms: Standard of Care

SUMMARY:
Problems with walking and balance are common in older adults with mild cognitive impairment. Walking and balance problems limit independence and increase risk for injuries due to falls. The purpose of this research study is to test the effectiveness of training that combines moving and thinking tasks, referred to as Personalized cognitive integrated sensorimotor virtual reality (VR)/mixed reality (MR) training on walking and balance ability. The study will also help to understand the changes in thinking ability and brain activity as a result of this training in older adults with mild cognitive impairment.

The study will evaluate the differences between two intervention groups (n=20 each): 1) personalized cognitive integrated sensorimotor VR/MR training (CM), and 3) standard of care (CTRL) on gait, balance, community ambulation, and cognitive functions, as well as underlying biomechanical and neurophysiological mechanisms to understand the changes due to CM.

ELIGIBILITY:
Inclusion Criteria:

* Between the age of 65 and 85 years for older adults.
* Montreal Cognitive Assessment (MOCA), 17 < MOCA < 24
* Medical clearance will be obtained from my clinician. If participants physician is unavailable the study team clinician will provide the medical clearance.
* Adequate cognitive function to give informed consent, understand the training and instructions, use the device and give adequate feedback.
* Able to stand for 5 minutes.

Exclusion Criteria:

* Body weight over 135 kgs.
* Uncontrolled or unstable seizure disorder.
* Severe joint contracture or spasticity of the ankle that limits passive range of motion as determined by the team.
* History of severe cardiac diseases such as myocardial infarction, coronary artery disease, cardiac arrhythmia, or congestive heart failure.
* Neuromuscular or neurological pathologies (e.g., spinal cord injury, stroke) that will interfere with ambulation.
* Uncontrolled or unstable orthostatic hypotension.
* Pre-existing conditions resulting in significant disruption in alignment or function of the lower limb during standing.
* History of injury or pathology to the lower limbs in the past 6 months or any medical issue precludes full weight-bearing and ambulation (e.g., orthopedic injuries).
* Diplopia or nystagmus.
* Walking speed from 10MWT >0.8m/s.

MRI specific exclusion criteria:

* Medications such as: steroids, benzodiazepines, and neuroleptics. The study doctor will review the medications with the participant.
* clip to repair a cerebral aneurysm (broken blood vessel in the head), cardiac pace-maker, cochlear implants (internal hearing aids) or metal fragments or pieces in the eyes or any other part of the body.
* non MRI compatible metal in any part of the body.
* Medical clearance from a physician that it is medically unsafe to receive regular MRI.
* Engage in the professions of painting or welding or other occupation that prevents me from getting a regular MRI.
* claustrophobia (fear of enclosed spaces).
* History of schizophrenia or bipolar disorder.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | 10 weeks
  TUG is a clinical test of functional gait abilities and dynamic balance. The participants will be asked to walk a distance of 3 meters from a seated position, turn around, walk back to the chair and sit back in the chair. The time taken to perform the task will be recorded using a stop watch. The TUG will be repeated multiple times. The participant may be asked to hold a plastic cup or count backwards by three from a randomly selected number while walking.
10 Meter walk test | 10 weeks
  Participants will be asked to walk about 12 meters. The time taken to walk 10 meters will be recorded.
Berg balance Assessment | 10 weeks
  This is a test that measures balance on a 5-point during routine tasks. The participant will be asked to perform 14 tasks involving: sitting, standing, reaching, lifting, and turning.
Fall Risk | 10 weeks
  The silver index will be measured using the Hunova (Movendo Srl., Italy) to quantify the risk of falls. The Silver Index tasks include static balance while eyes are open or closed, dynamic balance while standing on passive and elastic surfaces, limits of stability, reactive balance during perturbations, 6-meter walk, and sit-to-stand.
Balance | 10 weeks
  Root-mean-square of COM and COP displacements will be used to quantify balance tasks. COP will be obtained from Hunova. Whole body COM will be obtained using motion capture.
Temporal characteristics | 10 weeks
  This test assesses deviations in timing of steps during walking.
Spatial characteristics | 10 weeks
  This test assesses deviations in steplength during walking.
Physiological | 10 weeks
  The participants will wear small sensors on their body to assess the activity of the brain and muscles during walking and balancing tasks.
Digit Span (Wechsler Adult Intelligence Scale [WAIS-IV]) | 10 weeks
  This test assesses attention and working memory.
Flanker Inhibitory Control and Attention Test | 10 weeks
  This test assesses the allocation of limited attentional capacities to deal with an abundance of environmental stimulation. The test measures attention and the ability to inhibit response that may interfere with the ability to achieve goals.
Symbol Digit Modalities Test (SDMT) | 10 weeks
  This test assesses processing speed without a motor component
Paced Auditory Serial Addition Test (PASAT) | 10 weeks
  This test assesses information processing speed & ability and working memory
Letter-Number Sequencing (WAIS-IV) | 10 weeks
  This test assesses working memory
Delis-Kaplan Executive Function System | 10 weeks
  Selected subtests to assess executive function.
Community Ambulation | 10 weeks
  This test quantifies the amount of physical activity in the community using IMU sensors that participants will wear.
Continuous Performance Task | 10 weeks
  This test assesses attention.
Magnetic Resonance Imaging (MRI) | 1 week
  MRI scans will be performed to assess the structure and function of the brain while the participant is lying quietly in the MRI scanner.

SECONDARY OUTCOMES:
6 Minute Walk Test | 10 weeks
  Participants walk as far as possible for 6 minutes. They walk back and forth around the cones along an unobstructed pathway of 15 meters. They will be permitted to slow down or stop as necessary. The distance covered by the participant for the 6 minutes will be recorded at an interval of every 30 seconds using a measuring wheel and stop watch.
Dynamic Gait Index (DGI) | 10 weeks
  DGI is a measurement tool commonly used to assess dynamic balance, gait and risk for falls29. It consists of a total of eight gait assessments which can be scored on a four-point ordinal scale, ranging from 0-3, where '0' indicates the lowest level of function and '3' the highest level of function, allowing for a total possible score of 24.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Karunakaran, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No